CLINICAL TRIAL: NCT05836727
Title: Use of Laparoscopy in the Treatment of Pelvic Ring Ruptures
Acronym: PELVICOELIO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0010 - PELVICOELIO
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-02

CONDITIONS: Pelvic Fracture
Keywords: Pelvic ring surgery; Trauma Surgery; Plate Fixation; Laparoscopy; Case series
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Case series to describe the use of laparoscopy for the treatment of pelvic ring disruption.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent laparoscopy for the treatment of pelvic ring disruption

Exclusion Criteria:

* patient < 18 years old

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent laparoscopy for the treatment of pelvic ring disruption
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
conversion rate to open surgery | intraoperative
  conversion rate to open surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.